CLINICAL TRIAL: NCT03871660
Title: What Happens to Frequently Measured Glucose Measures in Patients, Both With and Without Diabetes, Who Are Receiving Total Parenteral Nutrition (TPN).
Brief Title: Flash Glucose Measurement in Patients on Total Parenteral Nutrition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LeedsNHS
Record Dates: First submitted 2019-02-21; First posted 2019-03-12 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus
Keywords: Total Parenteral Nutrition
MeSH Terms: conditions — Diabetes Mellitus; Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with diabetes on TPN (Other): Glucose levels will be monitored using the FreeStyle Libre devices over a 14 day period. In this time the patient will receive TPN.
  Interventions: Device: FreeStyle Libre Pro
- Patients without diabetes on TPN (Other): Glucose levels will be monitored using the FreeStyle Libre devices over a 14 day period. In this time the patient will receive TPN.
  Interventions: Device: FreeStyle Libre Pro

INTERVENTIONS:
Device: FreeStyle Libre Pro — Flash glucose monitoring device. Measures patients interstitial glucose levels continuously.

SUMMARY:
IV nutrition is a means of providing all the nutritional requirements of people who have severe bowel disease. At least 10% of people on longer term IV nutrition also have diabetes and IV nutrition includes delivering glucose directly to large veins. Unsurprisingly this causes elevated blood glucose levels, particularly in people with diabetes. This can make treatment of hyperglycaemia more challenging. As a result this study aims to use a flash glucose monitoring device, the FreeStyle Libre pro, to investigate what happens to glucose levels in patients receiving IV nutrition. We will look at this trend in 5 patients with diabetes and 5 patients without diabetes receiving IV nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Participants receiving TPN in Leeds with or without diabetes

Exclusion Criteria:

* Patients not receiving TPN
* Patients who do not speak English
* Patients who are unable to give consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Hyperglycaemia | 14 days
  Measurements of hyperglycaemia through interstitial glucose levels in patients on a TPN regime

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes, Endocrinology and General Medcine Department St James Hospital, Leeds, West Yorkshire, United Kingdom